CLINICAL TRIAL: NCT03408756
Title: A Randomized Controlled Trial Comparing the Efficacy and Safety Profile of Oral Versus Subcutaneous Route of Methotrexate Administration in Moderate to Severe Psoriasis
Brief Title: Comparison of Oral Versus Subcutaneous Route of Methotrexate Administration in Moderate to Severe Psoriasis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Dr. Tarun Narang, Assistant Professor of Dermatology, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: INT/IEC/2017/961
Record Dates: First submitted 2018-01-17; First posted 2018-01-24 (Actual); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Psoriasis Vulgaris
MeSH Terms: interventions — Methotrexate

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral Methotrexate (Active Comparator): Participants will receive methotrexate through oral route of administration
  Interventions: Drug: methotrexate
- Subcutaneous Methotrexate (Active Comparator): Participants will receive methotrexate through subcutaneous route of administration
  Interventions: Drug: methotrexate

INTERVENTIONS:
Drug: methotrexate — Participants will receive methotrexate through oral or subcutaneous route of administration
  Other Names: Folitrax; neotrexate

SUMMARY:
This study is a prospective, single blinded, randomized, pilot study to compare the effectiveness and safety profile of oral versus subcutaneous route of administration of methotrexate in management of patients with moderate to severe psoriasis. The recruited participants with moderate to severe psoriasis will be randomized into treatment arms. Randomization will be done using computer generated random number table. The participants in the first treatment arm will receive 0.3 mg/kg ( upto a maximum of 25 mg/week ) of weekly oral methotrexate for 12 weeks or achievement of PASI 90 whichever is earlier while the participants in second treatment arm will receive subcutaneous methotrexate at 0.3 mg/kg/week for the same duration. The participants will be followed at regular intervals and monitored adequately for hematological, hepatotoxic and other adverse effects both clinically and through laboratory investigations according to methotrexate consensus guidelines during the treatment period. PASI, percentage of body surface area (BSA) involvement and DLQI will be assessed at each follow up visit and at the end of 12 weeks. The treatment will be tapered at the rate of 5 mg/2 weeks and stopped after 12 weeks or achievement of PASI 90 whichever is earlier.. Follow ups will be done at every 2 weeks until treatment completion (12 weeks) and at every 4 weeks till 24 weeks after completion of treatment.

The primary outcome measures will be achievement of PASI 90 (90 % reduction in psoriasis area severity score (PASI) compared to baseline).The secondary outcomes will be improvement in DLQI (dermatology life quality index), relapse rate and adverse events if any.

DETAILED DESCRIPTION:
Introduction:

Methotrexate is one of the oldest and most commonly used systemic drugs for the treatment of psoriasis.[1] Even with the advent of other treatment modalities like systemic retinoids and biologics, methotrexate remains a popular modality for treatment of psoriasis owing to its cost-effectiveness, ease of administration and greater experience among practitioners regarding its use.[2] Despite long-term experience in the use of methotrexate in psoriasis, robust evidence and consensus regarding the ideal dosing schedule and route of administration is still lacking.[3] Oral route of methotrexate has been found to have unpredictable and non-linear bioavailability especially at doses greater than 15 mg/kg.[4] Subcutaneous route of methotrexate on the other hand is associated with better and more linear bioavailability at higher doses.4 Methotrexate by subcutaneous route has also been known to better tolerability and lesser gastrointestinal side effects as compared to oral route. [5] Recently conducted METOP study, which was a randomized controlled study comparing subcutaneous route of methotrexate administration and placebo in control of moderate to severe plaque psoriasis concluded that subcutaneous methotrexate is an efficient and safe modality of treatment of psoriasis. The study also suggested that the pace and longevity of response by subcutaneous route of methotrexate administration may be better than seen with oral route.[6] A recent retrospective study also concluded that subcutaneous route of methotrexate is an effective modality of treatment in patients of psoriasis who have failed oral methotrexate.[7] This study will be the first randomized controlled trial comparing oral versus subcutaneous route of administration of methotrexate in its efficacy in clearance of psoriasis and side effect profile. The study will help in clarification of dilemma of clinicians regarding the ideal route of administration of methotrexate in psoriasis. It will also further strengthen the evidence regarding the adverse effects and tolerability of subcutaneous route of methotrexate administration.

Methodology:

Aim of the study : To compare the effectiveness and safety profile of oral versus subcutaneous route of administration of methotrexate in patients with moderate to severe psoriasis.

This study will be an intention to treat single blinded randomized controlled trial. The participants will be patients with moderate to severe psoriasis fulfilling the inclusion and exclusion criteria . They will be randomly allocated to the two treatment arms in the beginning of the study. Participants in one treatment arm will receive methotrexate by oral route while participants in second treatment arm will receive methotrexate by subcutaneous route. Baseline PASI, percentage of body surface area involvement(BSA) and DLQI will be calculated for each patient at the start of study. Any systemic treatment will be stopped for a duration of at least 5 times their half lives before the start of methotrexate in each patient. The participants in first treatment arm will receive 0.3 mg/kg (upto a maximum of 25 mg/week ) of weekly oral methotrexate for 12 weeks or achievement of PASI 90 whichever is earlier while the patients in second treatment arm will receive subcutaneous methotrexate at 0.3 mg/kg/week for the same duration. The participants will be followed at regular intervals and monitored adequately for hematological, hepatotoxic and other adverse effects both clinically and through laboratory investigations according to methotrexate consensus guidelines during the treatment period. PASI, Body surface area (BSA) involvement and DLQI will be assessed at each follow up visit and at the end of 12 weeks. The treatment will be tapered at the rate of 5 mg/2 weeks and stopped after 12 weeks or achievement of PASI 90 whichever is earlier. The participants will be followed up for a period of 24 weeks after stopping methotrexate to observe the relapse free period.

Monitoring of the adverse effects:

Participants will be monitored for documented side effects of methotrexate at each follow up visit through history, clinical examination and laboratory investigations. The severity of adverse effects will be documented and decision regarding continuation and discontinuation of treatment will be taken as per the participant's will and guidelines.

Primary objectives

1. To compare the effectiveness of oral versus subcutaneous route of administration of methotrexate in patients with moderate to severe psoriasis.
2. To compare the safety profile of oral versus subcutaneous methotrexate.

Secondary objectives

1. Comparison between patients of both treatment arms with respect to time for achieving PASI 90 or PASI 100
2. Comparison between patients of both treatment arms in percentage of patients who achieve PASI 90 by the end of week 12 of treatment.
3. Comparison of improvement in DLQI between patients of both treatment arms.
4. Comparison of the relapse free period after stopping treatment.

Project schedule:

Screening and Patient recruitment: February 2018 to February 2019, Patient treatment and follow up: March 2018 to August 2018, Compilation of data: September 2019, Statistical analysis and Manuscript: October 2019.

Sample size and statistical analysis:

A total of 100 participants will be recruited in the study with 50 participants in each treatment arm. Independent -sample t-test will be used to compare group means in percentage decrease in PASI and percentage of patients developing adverse effects. Chi-square test will be used for qualitative variables. P value less than 0.05 will be considered significant.

Ethical Justification:

Informed consent will be obtained from each participant prior to recruitment in both the phases of study. Participants will be explained regarding both the arms of the study. The participants will have the right to withdraw without having to give reasons for doing so. Their refusal to participate in the study will not influence their future follow up with the institution in any way.

Methotrexate is the most commonly used systemic drug both in its oral and subcutaneous forms in the psoriasis clinic of investigator's institution and overall experience has suggested that it is an effective and safe drug. Monitoring of participants will be done by standard methotrexate consensus guidelines and treatment will be stopped if serious or intolerable adverse effects develop.

The investigators have also gathered sufficient experience regarding the efficacy and safety of subcutaneous route of methotrexate, especially in patients who have compliance issues or who have failed oral route or developed intolerable gastrointestinal adverse effects.

This study will be the first randomized controlled trial comparing oral versus subcutaneous route of administration of methotrexate in its efficacy in clearance of psoriasis and side effect profile. This study will help in clarification of dilemma of clinicians regarding the ideal route of administration of methotrexate in psoriasis with respect to effectiveness and tolerability. Subcutaneous route of methotrexate administration if found having better effectiveness and tolerability, can be tried first in patients who are failing or not tolerating oral methotrexate before switching to other modalities like retinoids and biologics. Subcutaneous methotrexate being cheaper than biologics and retinoids will also decrease the financial burden on psoriasis patients. Cost-effectiveness of subcutaneous methotrexate will be a major advantage for developing countries like India where most of the patients cannot afford retinoids or biologics. The ease of administration, availability and accessibility of subcutaneous methotrexate is also better than modalities like biologics and phototherapy in developing countries , especially in remote areas.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged more than 18 years with clinical diagnosis of plaque psoriasis
2. Patients with body surface area involvement > 10 %, PASI >10, DLQI >10.

Exclusion Criteria:

1. Hemoglobin < 8 gm/dl ,Total leukocyte count < 3500/ mm3, Platelet count < 100,000/mm3
2. Elevation of hepatic enzymes (alanine aminotransferase [ALT], aspartate aminotransferase [AST], or γ glutamyl transferase [GGT]) to more than twice the upper limit of normal.
3. Hepatitis, active or recurrent, cirrhosis or excessive current alcohol intake .
4. Use of other hepatotoxic drugs by the patient
5. Positive hepatitis B, hepatitis C or HIV serology
6. Pulmonary or extra-pulmonary active tuberculosis
7. Deranged renal function test.
8. Pregnancy or lactation or if patient is planning to conceive during the treatment period.
9. Patient on other immunosuppressive drugs
10. Recent live vaccination
11. Unreliable patient
12. Patients unwilling for monthly follow-ups. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-04-01 (Estimated); Primary Completion 2019-10-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
Achievement of PASI 90 | 12 weeks
  PASI 90 refers to 90 % reduction in psoriasis area severity score (PASI) compared to baseline

SECONDARY OUTCOMES:
Improvement in DLQI (dermatology life quality index) | 12 weeks
  Improvement in DLQI (dermatology life quality index) as compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Tarun Narang, MD, Principal Investigator — PGIMER Chandigarh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roenigk HH Jr, Auerbach R, Maibach H, Weinstein G, Lebwohl M. Methotrexate in psoriasis: consensus conference. J Am Acad Dermatol. 1998 Mar;38(3):478-85. doi: 10.1016/s0190-9622(98)70508-0. No abstract available. PMID 9520032
- [Background] Kalb RE, Strober B, Weinstein G, Lebwohl M. Methotrexate and psoriasis: 2009 National Psoriasis Foundation Consensus Conference. J Am Acad Dermatol. 2009 May;60(5):824-37. doi: 10.1016/j.jaad.2008.11.906. PMID 19389524
- [Background] Montaudie H, Sbidian E, Paul C, Maza A, Gallini A, Aractingi S, Aubin F, Bachelez H, Cribier B, Joly P, Jullien D, Le Maitre M, Misery L, Richard MA, Ortonne JP. Methotrexate in psoriasis: a systematic review of treatment modalities, incidence, risk factors and monitoring of liver toxicity. J Eur Acad Dermatol Venereol. 2011 May;25 Suppl 2:12-8. doi: 10.1111/j.1468-3083.2011.03991.x. PMID 21388454
- [Background] Schiff MH, Jaffe JS, Freundlich B. Head-to-head, randomised, crossover study of oral versus subcutaneous methotrexate in patients with rheumatoid arthritis: drug-exposure limitations of oral methotrexate at doses >/=15 mg may be overcome with subcutaneous administration. Ann Rheum Dis. 2014 Aug;73(8):1549-51. doi: 10.1136/annrheumdis-2014-205228. Epub 2014 Apr 12. PMID 24728329
- [Background] Bianchi G, Caporali R, Todoerti M, Mattana P. Methotrexate and Rheumatoid Arthritis: Current Evidence Regarding Subcutaneous Versus Oral Routes of Administration. Adv Ther. 2016 Mar;33(3):369-78. doi: 10.1007/s12325-016-0295-8. Epub 2016 Feb 4. PMID 26846283
- [Background] Warren RB, Mrowietz U, von Kiedrowski R, Niesmann J, Wilsmann-Theis D, Ghoreschi K, Zschocke I, Falk TM, Blodorn-Schlicht N, Reich K. An intensified dosing schedule of subcutaneous methotrexate in patients with moderate to severe plaque-type psoriasis (METOP): a 52 week, multicentre, randomised, double-blind, placebo-controlled, phase 3 trial. Lancet. 2017 Feb 4;389(10068):528-537. doi: 10.1016/S0140-6736(16)32127-4. Epub 2016 Dec 22. PMID 28012564
- [Background] Yesudian PD, Leman J, Balasubramaniam P, Macfarlane AW, Al-Niaimi F, Griffiths CE, Burden AD, Warren RB. Effectiveness of Subcutaneous Methotrexate in Chronic Plaque Psoriasis. J Drugs Dermatol. 2016 Mar;15(3):345-9. PMID 26954320